CLINICAL TRIAL: NCT07234084
Title: The Effectiveness of Functional Magnetic Stimulation in the Physiotherapeutic Rehabilitation of Athletes With Bone Marrow Edema: A Randomized Controlled Trial
Brief Title: Functional Magnetic Stimulation (FMS) for Bone Marrow Edema in Athletes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Hellenic University (Other)
Responsible Party: Principal Investigator, Dimitrios Lytras, Assistant Professor of Physiotherapy, International Hellenic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC-15/2025
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Bone Marrow Edema
Keywords: Bone Stress Injury; Functional Magnetic Stimulation; Physiotherapy; Rehabilitation

STUDY DESIGN:
Intervention Model Description: A single-assessor-blind randomized controlled trial lasting four weeks, with a twelve-week follow-up, will be conducted on forty athletes diagnosed with MRI-confirmed bone marrow edema of the lower limb graded as Fredericson 2 or 3. Participants will be randomly allocated into two groups of twenty each (intervention and control). The intervention group will receive a combined treatment consisting of a standardized physiotherapy rehabilitation program and Functional Magnetic Stimulation (two sessions per week for four weeks), while the control group will follow the same physiotherapy protocol without FMS. Clinical assessments of pain and functional ability will be performed at baseline, at two weeks, at the end of the four-week intervention, and at sixteen weeks to monitor short- and medium-term recovery. MRI will be conducted at baseline, week 4, and week 16 to document radiological changes in bone marrow edema.
Who Masked: Outcomes Assessor
Masking Description: A masked assessor will conduct the measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapy plus Functional Magnetic Stimulation (FMS) (Experimental): Participants allocated to this group will receive 12 sessions of a conventional physiotherapy protocol and 8 sessions of FMS.
  Interventions: Other: Conventional Physiotherapy with FMS
- Physiotherapy without Functional Magnetic Stimulation (FMS) (Active Comparator): Participants allocated to this group will receive 12 sessions of a conventional physiotherapy protocol without the FMS
  Interventions: Other: Conventional Physiotherapy without FMS

INTERVENTIONS:
Other: Conventional Physiotherapy with FMS — Participants will receive a standardized four-week physiotherapy program, three sessions per week (12 sessions in total), each lasting approximately 45 minutes. Treatment will include therapeutic exercise for progressive strengthening and flexibility, manual therapy for pain modulation, and unloading-reloading strategies to restore functional load tolerance. Exercises will be tailored to the recovery stage, and participants will be instructed on home exercises and activity modification.
  In addition, participants will receive Functional Magnetic Stimulation (FMS) twice weekly for four weeks (eight sessions in total). Each session will last 30 minutes. FMS will be applied directly over the affected region using a fixed frequency of 40 Hz without modulation. The stimulation duty cycle will consist of an active phase of 3 seconds followed by a rest period of 6 seconds. Intensity will be gradually adjusted to patient tolerance avoding scomfort or excessive contraction.
  Arms: Physiotherapy plus Functional Magnetic Stimulation (FMS)
Other: Conventional Physiotherapy without FMS — Participants in this group will follow the same conventional physiotherapy protocol as the first group, without the application of FMS
  Arms: Physiotherapy without Functional Magnetic Stimulation (FMS)

SUMMARY:
This randomized controlled trial investigates the effectiveness of Functional Magnetic Stimulation (FMS) as an adjunct to physiotherapy in athletes with MRI-confirmed bone marrow edema of the lower limb. Forty athletes with Fredericson grade 2-3 edema will be randomly assigned to receive either physiotherapy plus FMS or physiotherapy alone for four weeks. Clinical, functional, and imaging assessments will be conducted up to 16 weeks. Primary outcomes include pain intensity, lower-limb function, return-to-sport readiness, and MRI indicators of bone marrow edema. The study aims to determine whether adjunctive FMS enhances recovery and accelerates the resolution of bone marrow edema compared with standard physiotherapy.

DETAILED DESCRIPTION:
Background: Bone marrow edema is a reversible stress-related bone injury in athletes, causing localized pain during loading and confirmed by MRI, the gold standard for diagnosis and monitoring. Grades 2 and 3 of the Fredericson classification represent clinically significant edema without a fracture line and are managed conservatively through physiotherapy including exercise, manual techniques, and gradual reloading. Functional Magnetic Stimulation (FMS) is a non-invasive method that induces deep neuromuscular activation and improves circulation. Although increasingly used in musculoskeletal rehabilitation, its effect on recovery from bone marrow edema has not yet been tested in a controlled clinical setting.

Aim: The aim of the present randomized controlled clinical trial is to evaluate the effectiveness of adding Functional Magnetic Stimulation to a structured physiotherapy rehabilitation program in athletes with MRI-confirmed bone marrow edema of the lower limb. The primary objective is to determine whether the combined approach results in greater clinical improvement, superior functional recovery, and faster radiological resolution of edema compared with physiotherapy alone.

Method: Forty athletes with lower-limb bone marrow edema graded as Fredericson 2 or 3 on MRI will be randomly assigned to two groups. The intervention group will follow a four-week physiotherapy program combining therapeutic exercise, manual therapy, and unloading techniques with Functional Magnetic Stimulation applied twice weekly. The control group will receive the same physiotherapy without FMS. Assessments will occur at baseline, two, four, and sixteen weeks, including pain (NRS 0-10), functional ability (LEFS-GR), and readiness for return to sport (Tegner scale). MRI at baseline, week 4, and week 16 will evaluate Fredericson grade, edema intensity, and edema extent. All parameters are predefined as primary outcomes. Data will be analyzed with mixed-model ANOVA for repeated measures with the significance level set at p < .05.

Expected Results: It is anticipated that athletes receiving Functional Magnetic Stimulation in addition to physiotherapy will show greater pain reduction, improved lower-limb function, faster MRI-documented resolution of bone marrow edema, and earlier readiness to return to sport compared with physiotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Athletes aged 18-45 years participating in regular sports training ≥3 sessions per week for the past 6 months.
* MRI-confirmed bone marrow edema (BME) of the lower limb graded as Fredericson 2 or 3.
* Onset of pain or symptoms within the previous 6 weeks.
* Pain intensity ≥4/10 on the Numeric Rating Scale during loading activity.
* Ability to comply with the 4-week intervention and 16-week follow-up assessments.
* Written informed consent provided prior to participation.

Exclusion Criteria:

* Fredericson grade 4 or evidence of a fracture line on MRI. Bone marrow edema secondary to infection, tumor, or systemic inflammatory disease.
* History of recent fracture, surgery, or intra-articular injection in the affected limb within 12 weeks.
* Prior exposure to Functional Magnetic Stimulation or Extracorporeal Shockwave Therapy within 8 weeks before enrollment.
* Presence of metallic implants, pacemaker, or other contraindications to magnetic stimulation.

Pregnancy or breastfeeding. Use of systemic corticosteroids or medications affecting bone metabolism. Any neurological, metabolic, or cardiovascular condition interfering with safe participation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Changes in pain intensity with Numeric Rating Scale (NPRS) | pre-treatment, week 4, Week 16
  This tool is an eleven-point pain scale numbered from zero to 10. The left end of the scale corresponds to zero and is marked as "No pain", whereas the right end corresponds to 10 and is marked as "Maximum pain". Consequently, a higher value indicates more intense pain (Childs et al, 2005). The examinee is asked to choose an integer that best reflects the intensity of their pain. Participants will be asked to rate their pain under three conditions: at rest, during standardized loading of the affected limb, and during hypothetical return to sport.The NPRS is widely used to measure pain in both clinical practice and research, showing high test-retest reliability and high conceptual construct validity.
Changes in lower-limb functional ability with the Greek Version of the Lower Extremity Functional Scale (LEFS-GR) | baseline, week 4, week 16
  The LEFS-GR is a self-reported questionnaire consisting of 20 items that assess the degree of difficulty in performing everyday and sport-related lower-limb activities. Each item is rated on a 5-point scale (0 = extreme difficulty or unable to perform; 4 = no difficulty), yielding a total score from 0 to 80, with higher scores indicating better functional ability. The Greek version of the LEFS has demonstrated excellent internal consistency (Cronbach's α = 0.974) and test-retest reliability (ICC = 0.986, p < 0.001) in individuals with lower-limb musculoskeletal disorders (Stasi et al., 2012).
Changes in bone marrow edema characteristics with Magnetic Resonance Imaging (MRI) | baseline, week 4, week 16
  Magnetic Resonance Imaging (MRI) will be used to evaluate changes in bone marrow edema (BME) according to the Fredericson classification, which grades stress-related bone injury from 0 (normal) to 4 (cortical fracture). MRI scans will include T1-weighted and fat-suppressed T2/STIR sequences obtained under identical imaging parameters at all time points. Semi-quantitative analysis will be performed to record (a) Fredericson grade, (b) bone marrow edema signal intensity on a 0-3 scale, and (c) edema extent as a percentage of the total bone volume.
Changes in return-to-sport readiness with the Tegner Activity Scale and perceived sport pain | baseline, week 4, week 16
  The Tegner Activity Scale (TAS) is an 11-level ordinal scale designed to evaluate physical activity and sports participation following lower-limb injury. It ranges from 0 (inability to work or perform daily activities due to symptoms) to 10 (participation in competitive sports at national or elite level). The validated Greek version (Gr-TAS) demonstrates high internal consistency (Cronbach's α = 0.89) and test-retest reliability (ICC = 0.97) in musculoskeletal populations (Panagopoulos et al., 2020). In this study, the scale will be combined with a perceived sport-related pain score (NRS 0-10), where higher TAS scores and lower pain scores will indicate greater readiness to return to sport.

CONTACTS AND LOCATIONS:
Overall Officials: Paris Iakovidis, PhD, Study Chair — International Hellenic University
Locations (1):
- Department of Physiotherapy, Faculty of Health Sciences International Hellenic University, Thessaloniki, Sindos, Greece

IPD SHARING:
Plan to Share IPD: No